CLINICAL TRIAL: NCT00210717
Title: A Randomized, Double-Blind, Parallel Group, Comparative Study of Flexibly Dosed Paliperidone Palmitate (25, 50, 75, or 100 mg eq.) Administered Every 4 Weeks and Flexibly Dosed RISPERDAL CONSTA (25, 37.5, or 50 mg) Administered Every 2 Weeks in Subjects With Schizophrenia
Brief Title: A Study to Compare the Effectiveness and Safety of Flexibly Varied Doses of Paliperidone Palmitate and Risperidone in Treating Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004195
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia
Keywords: schizophrenia; intramuscular injection; antipsychotic agents; risperidone; paliperidone palmitate; dementia praecox; mental disorders; PANSS
MeSH Terms: conditions — Schizophrenia; Mental Disorders | interventions — Paliperidone Palmitate

INTERVENTIONS:
Drug: paliperidone palmitate

SUMMARY:
The purpose of this study is to compare the effectiveness and safety over 1 year of treatment of intramuscular injections of paliperidone palmitate and long-acting risperidone in patients with schizophrenia.

DETAILED DESCRIPTION:
Paliperidone palmitate is being developed as a long-acting intramuscular injectable formulation for the treatment of schizophrenia. Many patients with schizophrenia achieve symptom stability with the available oral antipsychotic medications; however, it is estimated that up to 75% have difficulty adhering to a daily oral treatment regimen. Long-acting injectable formulations may make compliance with the treatment regimen easier by eliminating the need for daily medication. An injectable formulation of risperidone is widely used in the treatment of schizophrenia and has been well tolerated by patients with chronic schizophrenia at the recommended dosage of 25 to 50 milligrams every 2 weeks. The present study is designed to evaluate the comparability of paliperidone palmitate and long-acting injectable risperidone over 1 year of treatment.

This is a randomized, double-blind, active-controlled, parallel-group, multicenter comparative study in patients with schizophrenia. The study comprises a screening period of up to 1 week (including periods for washout of psychotropic medications and, if necessary, an oral tolerability test) and a 53-week double-blind treatment period. In the double-blind treatment period, patients will be randomly assigned in equal numbers to receive treatment with either (1) flexibly dosed paliperidone palmitate administered every 4 weeks or (2) flexibly dosed long-acting risperidone administered every 2 weeks. Drug effectiveness and safety will be evaluated periodically throughout the study. Samples for pharmacokinetic evaluation will be collected at designated time points, and a blood sample will be collected at baseline (before the start of the double-blind treatment period) or at any subsequent visit for an optional pharmacogenomic (genetic) analysis. The study hypothesis is that paliperidone palmitate will be as effective as long-acting risperidone in the treatment of patients with schizophrenia. Paliperidone palmitate (25, 50, 75, or 100 milligrams (mg) equivalent) every 4 weeks, or long-acting risperidone 25, 37.5, or 50 mg every 2 weeks of double-blind treatment period, injected into the gluteal muscle (buttocks). Oral risperidone (1-6 mg) first 4 weeks of double-blind period

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of schizophrenia (disorganized, catatonic, paranoid, residual, or undifferentiated types) according to the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM IV) for at least 1 year before the screening evaluation
* a total PANSS score of 60 to 120 at screening and baseline (pre-treatment) evaluations
* a body mass index (BMI [weight (kilograms)]/[height (meters)]²) of at least 15.0 kg/m² .

Exclusion Criteria:

* A primary active DSM-IV Axis I diagnosis other than schizophrenia
* a decrease of 25% or more in the total PANSS score between screening and baseline evaluations
* a DSM-IV diagnosis of active substance dependence within 3 months of screening evaluation
* a history of treatment resistance as defined by failure to respond to 2 adequate trials of different antipsychotic medications
* a woman who is pregnant, breast-feeding, or planning to become pregnant during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 748 (Actual)
Dates: Start 2005-02; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
The change in the total score of the Positive and Negative Syndrome Scale (PANSS) from the beginning to the end of the double-blind treatment period or to the last post-randomization assessment.

SECONDARY OUTCOMES:
The investigator's Clinical Global Impression of the Severity (CGI-S) of schizophrenia and rating of mental function on a Personal and Social Performance Scale (PSP). Evaluations of adverse events, laboratory tests, and other measures of drug safety.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Fleischhacker WW, Gopal S, Lane R, Gassmann-Mayer C, Lim P, Hough D, Remmerie B, Eerdekens M. A randomized trial of paliperidone palmitate and risperidone long-acting injectable in schizophrenia. Int J Neuropsychopharmacol. 2012 Feb;15(1):107-18. doi: 10.1017/S1461145711001076. Epub 2011 Jul 22. PMID 21777507
- See also: A study to compare the efficacy and safety of flexibly varied doses of paliperidone palmitate and risperidone in treating patients with schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=563&filename=CR004195_CSR.pdf